CLINICAL TRIAL: NCT05240885
Title: Metabolic and Functional Consequences of Aging in Health and Disease
Status: Recruiting | Type: Observational
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Professor & Chancellor Edges Fellow, Texas A&M University
Other Study IDs: 2021-1413; 82-Aging (Other: CTRAL)
Record Dates: First submitted 2022-01-19; First posted 2022-02-15 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Aging
Keywords: stable isotopes; disease; metabolism
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Controls: Study subjects that are eligible based on inclusion/exclusion criteria
  Screening visit: body weight and composition by DXA, height, and vital signs will be assessed.
  Study day(s): may include combinations of stable tracer infusions and with blood draws, cognitive and muscle performance testing
  Interventions: Other: Stable tracer infusion in a postabsorptive state

INTERVENTIONS:
Other: Stable tracer infusion in a postabsorptive state — Multiple stable-labeled tracers of amino acids, ketoacids, glycerol, short-chain fatty acids
  Other Names: Stable tracer infusion

SUMMARY:
Considerable heterogeneity in the aging population has been observed. The exceptional longevity of individuals reaching 100 years old, so-called centenarians may be an example of life-long healthy aging, or added years may be spent in poor health with decreased physical and cognitive functioning. Current knowledge of the aging experience and the trajectories of physical and cognitive decline across various age groups are not well-understood, yet crucial to prevent spending added years in disease. Hence, the study objective is to develop the metabolic profile associated with aging-related disorders measured as the incidence of impaired functional capacity, cognitive function, and/or well-being.

DETAILED DESCRIPTION:
Our lab developed a pulse method combining multiple stable tracers to study multiple metabolic pathways in the same individual simultaneously. By measuring whole-body metabolism in a large group of older adults, we may be able to unravel age-related deterioration in protein turnover (synthesis and breakdown) that contributes to impaired functional capacity. Metabolic profiles could explain differences in pathways in the aging process with a special interest in the metabolism of amino acids as they have been associated with aging-related disorders. Studies on the effect of aging on metabolism might serve as potential therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Stable body-weight (± 5%) for the past 3 months
* Subject is judged to be in satisfactory health based on medical history, physical examination, and laboratory screening evaluations.
* Ability to walk, sit down and stand up independently or with walking mobility aids
* Ability to lie in a supine or elevated position for up to 3 hours
* Willingness and ability to comply with the protocol

Exclusion Criteria:

* Insulin dependent diabetes mellitus
* Established diagnosis of malignancy
* History of untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Presence of fever within the last 3 days
* Use of short course of oral corticosteroids within 4 weeks preceding study day
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* (Possible) pregnancy
* Already enrolled in another clinical trial and that clinical trial interferes with participating in this study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will screen 200 subjects (to complete n=100). This number includes screen failures and drop-outs. We expect some dropout between screening and enrollment. Subjects who drop out prior to the successful completion of the study will be replaced. Data will be used up to the point of withdrawal. Age range: 50 years or older, inclusive; Ethnicity: all races and ethnicities.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Age-related changes in whole-body protein and amino acid metabolism | 2 hours
  Whole-body production rate measured after stable tracer administration

SECONDARY OUTCOMES:
Age-related changes in whole-body glucose metabolism | 2 hours
  Whole-body production rate measured after stable tracer administration
Age-related changes in whole-body fat metabolism | 2 hours
  Whole-body production rate measured after stable tracer administration
Age-related changes in depression as measured by the Hospital Anxiety and Depression Scale (HADS) and Geriatric Depression Scale (if applicable) | baseline visit
  Self-reported depression measured by a validated questionnaire related to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms). A higher score indicates a worse outcome (greater self-reported depression symptoms).
Age-related changes in anxiety as measured by the Hospital Anxiety and Depression Scale (HADS) | baseline visit
  Anxiety measured by a validated questionnaire related to anxiety-related symptoms. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) related to anxiety. A higher score indicates a worse outcome (greater self-reported anxiety symptoms).
Age-related changes in mood as measured by the Profile of Mood State (POMS) | baseline visit
  A psychological distress scale to measure the mood disturbance in 6 domains - fatigue-inertia, vigor-activity, tension-anxiety, depression-dejection, anger-hostility, and confusion-bewilderment in the past week. Each item on the questionnaire is awarded a score from 0 ("not at all") to 4 ("extremely"), except "Relaxed" and "Efficient" scored 4 ("not at all") and 0 ("extremely"), based on the intensity of the assessed feeling in the past week.
Age-related changes in health status | baseline visit
  Health status assessed by Health-Related Quality of Life Scale (HR-QoL)
Age-related changes in physical activity | baseline visit
  Physical activity assessed by Physical Activity Scale for the Elderly (PASE)
Age-related changes in sleep quality | baseline visit
  Sleep quality assessed by Pittsburgh Sleep Quality Index
Age-related changes in nutritional status | baseline visit
  Nutritional status assessed by Mini-Nutritional Assessment
Age-related changes in attention and executive functions as measured by Trail Making Test (TMT) | baseline visit
  In Part A, the examinee is instructed to connect a set of 25 circles with numbers as quickly as possible while maintaining accuracy. In Part B, the examinee is instructed to connect a set of 25 circles, alternating between numbers and letters, as quickly as possible while maintaining accuracy. Measures attentional resources and is a measure of the frontal lobe "executive" functions of visual search, set-switching and mental flexibility. The total time in seconds was reported for each measure.
Age-related changes in overall cognitive abilities as measured by Montreal Cognitive Assessment (MoCA) | baseline visit
  MoCa assesses several cognitive domains and is used for the screening of mild cognitive impairment. Total scores range from 0-30 with lower scores indicating decreased functioning.
Age-related changes in exercise capacity | baseline visit
  Functional exercise capacity assessed by 6-minute walk test
Age-related changes in physical weakness (frailty) | baseline visit
  Physical weakness assessed by Short Physical Performance Battery
Age-related changes in skeletal muscle strength of the upper extremity | baseline visit
  Skeletal muscle strength measured by handgrip test
Age-related changes in skeletal muscle strength of the lower extremity | baseline visit
  Skeletal muscle strength measured by one-leg test
Age-related changes in respiratory muscle strength | baseline visit
  Respiratory muscle strength measured by a hand-held mouth pressure device (Micro RPM)
Age-related changes in balance | baseline visit
  Skeletal muscle strength measured by Berg Balance Scale and balance platform
Age-related changes in gut microbiota | baseline visit
  The amount and types of microbiota assessed in collected stool sample
Age-related changes in gut function | baseline visit
  Gut function assessed by Gastrointestinal Symptom Rating Scale, a 15-item instrument designed to assess the symptoms associated with common gastrointestinal disorders. A higher score indicates worse outcomes (more discomfort).

OTHER OUTCOMES:
Age-related changes in hand dexterity | baseline visit
  Hand dexterity assessed by the Nine-Hole Peg Test (9-HPT), a standardized, quantitative assessment in which the subject is asked to take pegs from a container, one by one, and place them into the holes on the board. Time upon completion will be recorded using both left and right hand, separately.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Clinical Research Building, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared upon request for up to 6 years beyond completion of the trial based on methods/proposal approved by both parties' institutional review committees. Individual participant data that underlie the results of the trial may be shared after de-identification (text, tables, figures, and appendices). Additional documents available per request include: study protocol, statistical analysis plan, and informed consent. Requests should be directed to Dr. Marielle Engelen (mpkj.engelen@ctral.org).